CLINICAL TRIAL: NCT03897023
Title: Anaylsis of Gut Microbiota in ICU
Brief Title: Gut Microbiota Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Maru Kim, Assistant Professor, The Catholic University of Korea
Other Study IDs: GMPS1
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Microbiota; Metabolism
MeSH Terms: interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stable patient: Stable patients who admitted to ICU for observation.
  Interventions: Biological: Gut Microbiota

INTERVENTIONS:
Biological: Gut Microbiota — Status of microbiota

SUMMARY:
Microbiota is known to effect metabolism. This is pilot study to get status of microbiota from normal control. It will be compared to data from specific patients in ICU via further study.

DETAILED DESCRIPTION:
Microbiota is known to effect metabolism. This is pilot study to get status of microbiota from normal control. It will be compared to data from specific patients in ICU via further study.

ELIGIBILITY:
Inclusion Criteria:

* Older than 17 years old
* Every patients who are admitted to ICU

Exclusion Criteria:

* With history of disease such as cancer, Crohn's disease, ulcerative colitis, irritable bowel syndrome
* With history of immunosuppressive agents.
* Initial systolic blood pressure <100
* Initial pulse rate > 100
* Need emergent operation at brain or torso
* Need vasopressor, transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable adult patient who are admitted to ICU
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-06-27 (Estimated); Study Completion 2021-06-27 (Estimated)

PRIMARY OUTCOMES:
Stuatus of gut microbiota in stable patient | 1 Month
  Result of next generation sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Uijeongbu St.Mary's hospital, Uijeongbu-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No